CLINICAL TRIAL: NCT07004452
Title: Multi-modal Adverse Events Prediction for Premature Coronary Heart Disease Trial: MAP-CHD Trial
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023ZD0504003
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Premature Coronary Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational cohort study is to establish a risk prediction model for adverse events in Chinese individuals under 45 years old with premature coronary artery disease. The main questions it aims to answer are:

* What are the major risk factors for poor prognosis in Chinese patients with premature coronary artery disease?
* What is the difference in the prognosis of patients with premature coronary heart disease with different phenotypes? Participants taking no mandatory intervention will be followed up for 2 year, with blood tests at 1 year and outpatient or telephone interviews at other timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years;
* Clinically confirmed CAD with ≥50% luminal stenosis in at least one major coronary artery or significant branch, verified by coronary angiography;
* For acute coronary syndrome (ACS) or percutaneous coronary intervention (PCI) patients: clinical stability meeting discharge criteria post-treatment;
* Voluntary participation with signed informed consent.

Exclusion Criteria:

* Heart transplant recipients;
* Severe systemic comorbidities with life expectancy <1 year;
* Previous enrollment in other drug/device clinical trials without completing the primary endpoint observation period;
* Inability to comply with follow-up (e.g., dementia, severe psychiatric disorders).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Eligible participants are CAD patients aged 18-45 years confirmed by coronary angiography or other imaging modalities, including those with stable/unstable angina or myocardial infarction.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
MACCE, defined as a composite of cardiac death, MI, ischemic stroke, and repeat revascularization | 2 years
Sensitivity for 2-year MACCE prediction | 2 years
  For the validation cohort
Specificity for 2-year MACCE prediction | 2 years
  For the validation cohort

SECONDARY OUTCOMES:
Incidence of death (cardiovascular, noncardiovascular, and undetermined) at 1 m, 6 m, 1 y and 2 y | 2 years
  For the development cohort
Incidence of MI (target vessel related and non-target vessel related or Culprit and non-culprit lesion-related) at 1 m, 6 m, 1 y and 2 y | 2 years
  For the development cohort
Incidence of all revascularizations (ischemia driven vs. non-ischemia driven; Target vs. non-target vessel; Culprit vs. non-culprit lesion) at 1 m, 6 m, 1 y and 2 y | 2 years
  For the development cohort
Incidence of definite or probable stent thrombosis during the acute, subacute, late, and very late phase according to the ARC-2 criteria | 2 years
  For the development cohort
Incidence of stroke (ischemic and hemorrhagic stroke) at 1 m, 6 m, 1 y and 2 y | 2 years
  For the development cohort
Incidence of bleeding events defined as BARC type ≥2 at 1 m, 6 m, 1 y and 2 y | 2 years
  For the development cohort
Area under the ROC curve (AUC) | 2 years
  For the validation cohort
Positive predictive value (PPV) | 2 years
  For the validation cohort
Negative predictive value (NPV) | 2 years
  For the validation cohort

CONTACTS AND LOCATIONS:
Locations (1):
- FuWai Hospital, Beijing, China